CLINICAL TRIAL: NCT05246436
Title: Effect of Warm Fluid Distension Media in Relieving Pain in Outpatient Hysteroscopy: Randomized Controlled Trial.
Brief Title: Effect of Warm Fluid Distension Media in Relieving Pain in Outpatient Hysteroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amira Mohamed (Other)
Responsible Party: Sponsor-Investigator, Amira Mohamed, principal investigator, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FMASU MS 567/2021
Record Dates: First submitted 2022-01-12; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Office Hysteroscopy
Keywords: warm saline

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- warm saline (Active Comparator): Patients who used warm saline as a distention media in office hysteroscopy
  Interventions: Procedure: warming saline media
- room temperature saline (Sham Comparator): Patients who used room temprature saline as a distention media in office hysteroscopy
  Interventions: Procedure: room temperature saline media

INTERVENTIONS:
Procedure: warming saline media — use warm saline as a distention media in office hysteroscopy
  Arms: warm saline
Procedure: room temperature saline media — use room temperature saline as a distention media in office hysteroscopy
  Arms: room temperature saline

SUMMARY:
The aim of study is to determine if the use of warm saline distention media during outpatient hysteroscopy reduces Pain/discomfort of the procedure.

Research hypothesis: In women undergoing office hysteroscopy, there will be reduced pain perception when using warm saline (body temperature 37°C during office hysteroscopy.

Research question: In women undergoing office hysteroscopy, Will there be a difference in pain perceived during the procedure if the investigators use warm saline(body temperature 37°C) rather than normal saline (room temperature) as a distension media?

DETAILED DESCRIPTION:
Office hysteroscopy is a procedure where a doctor uses a thin tube with a tiny camera to look inside the uterus. There are no incisions. Saline solution is used to expand the uterus in order to look at the inside of the uterus .

The vaginoscopic 'non-touch' technique first described by Bettocchi and Selvaggi (1997) has avoided the need for using a speculum and tenaculum in outpatient hysteroscopy; miniaturization of fibreoptic instruments has also enabled the procedure to be conducted without intra- or paracervical anesthesia.

Indications for diagnostic & therapeutic outpatient hysteroscopy include abnormal uterine bleeding, reproductive problems, glandular abnormalities on cervical smear, identification and retrieval of lost intrauterine devices, polypectomy, endometrial ablation and myomectomy.

Hysteroscopic procedures can be successfully performed in an office setting without any anesthesia.

There are pharmacological and non pharmacological analgesic methods. Non pharmacological methods, such as vaginoscopy or mini hysteroscopes, are advisable to avoid producing pain . The pharmacological method including intervention method which is para cervical block, reducing pain during and 30 minutes after hysteroscopy. And medical methods such as Non steroidal anti-inflammatory drugs (NSAIDs) seem to be useful in the postoperative period. Evidence is not clear about combination of techniques or misoprostol .

Endometrial cavity is an empty cavity and requires distension to permit visualization. Therefore, during hysteroscopy either fluid or carbon dioxide gas is used to enlarge the endometrial cavity. To achieve a panoramic view, the uterine walls must be forcibly separated. The thick muscle of uterine walls needs a minimum pressure of 40 mm Hg to distend the cavity adequately for hysteroscopic visualization.

Normal saline is usually recommended as the distention medium in outpatient hysteroscopy as it allows improved image resolution and is associated with less vasovagal episodes compared with carbon dioxide. Although it is thought that uterine contractility could be provoked by instillation of saline at lower temperatures, there is little data on the effect of temperature on clarity of image, discomfort/pain, outcome of the procedure and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* - Age ≥ 18 years old.
* Indications of diagnostic hysteroscopy: Cases complaining of abnormal uterine bleeding and /or undergoing the procedure to assess the endocervical canal, uterine cavity, and tubal Ostia for infertility, removal of foreign body, Suspected Mullerian anomalies.

Exclusion Criteria:

* - Contra-indications of diagnostic hysteroscopy: unable to exclude pregnancy, acute pelvic infection, active genital herpes, confirmed cervical or endometrial cancer and profuse bleeding at the time of the procedure.
* Any usage of analgesic agent on the day of the procedure.
* Failure of entry of the cervical canal requiring cervical dilatation.
* Any additional procedure during the procedure: polypectomy, biopsy and adhesiolysis.
* Patient refusal to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
warm saline versus room temp. saline as a distention media in office hysteroscopy in reliving pain by usage of the visual analog scale (VAS) | base line
  The patient makes a mark on the visual analog scale line to indicate the intensity of her pain. Pain will be measured using a 10-cm visual analogue scale (VAS) graded from 0 to 10 , (0) means no pain (better outcome), and (10) means worst possible pain (worse outcome)

SECONDARY OUTCOMES:
The clarity of the view.(questionnaire). | base line
  questionnaire including clear (better outcome) or dim (worse out come)

OTHER OUTCOMES:
The ease of entry of the hysteroscopy.(questionnaire) | base line
  questionnaire including easy (better out come) difficult (worse out come)
Patient satisfaction.(questionnaire) | base line
  questionnaire including yes (better outcome ) No (worse outcome)
Time of the procedure.(time by minutes) | base line
  calculate time of each procedure by minutes
complications (questionnaire) | base line
  questionnaire including No complications ( better outcome ) complications happen (worse outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospital, Cairo, Egypt

REFERENCES:
- [Background] Issat T, Beta J, Nowicka MA, Durczynski A, Jakimiuk AJ. Pain assessment during outpatient hysteroscopy using room temperature versus warm normal saline solution as a distention medium - a prospective randomized study. Clin Exp Obstet Gynecol. 2017;44(3):359-363. PMID 29949273